CLINICAL TRIAL: NCT00624962
Title: Pilot Study of Early Enteral Tube Feedings in Children Receiving Chemotherapy for Newly Diagnosed AML/MDS and High Risk Solid Tumors
Brief Title: Early Enteral Tube Feedings in Children Receiving Chemo for AML/MDS & High Risk Solid Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John B. Pietsch, Associate Professor of Pediatric Surgery and Pediatrics, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000583517; VU-VICC-PED-0604; VU-VICC-060151
Record Dates: First submitted 2008-02-27; First posted 2008-02-28 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2010-11

CONDITIONS: Brain and Central Nervous System Tumors; Kidney Cancer; Leukemia; Liver Cancer; Neuroblastoma; Sarcoma; Solid Tumor
Keywords: childhood soft tissue sarcoma; neuroblastoma; childhood hepatoblastoma; childhood cerebellar astrocytoma; childhood ependymoma; childhood brain stem glioma; childhood meningioma; childhood myelodysplastic syndromes; unspecified childhood solid tumor, protocol specific; childhood acute myeloid leukemia/other myeloid malignancies; central nervous system neoplasm; Wilms tumor and other childhood kidney tumors; childhood brain tumor; childhood medulloblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Kidney Neoplasms; Leukemia; Liver Neoplasms; Neuroblastoma; Sarcoma; Hepatoblastoma; Familial ependymoma; Meningioma; Wilms Tumor; Medulloblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Correlative/Supportive Care (Other)
  Interventions: Dietary Supplement: nutritional intervention; Dietary Supplement: therapeutic nutritional supplementation

INTERVENTIONS:
Dietary Supplement: nutritional intervention — Nutritional status assessment on enrollment in study, beginning of course 1 and end of study period (week 12 or beginning of Course 5 chemotherapy)
  Other Names: Non indicated
Dietary Supplement: therapeutic nutritional supplementation — enteral feedings via a nasogastric tube for 50% or more of the total nutritional support days.
  Other Names: not indicated

SUMMARY:
RATIONALE: Tubefeeding may help maintain good nutrition and lessen weight loss in younger patients receiving chemotherapy for cancer.

PURPOSE: This clinical trial is studying how well tube feedings work in younger patients receiving chemotherapy for newly diagnosed acute myeloid leukemia, myelodysplastic syndrome, or high-risk solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the feasibility and acceptance of undertaking early enteral tube feedings in children receiving induction chemotherapy for newly diagnosed acute myeloid leukemia or myelodysplastic syndromes, primary cancers of the central nervous system, or high-risk solid tumors.

Secondary

* To determine the safety of proactive enteral nutrition in these patients.
* To evaluate the effect of enteral nutrition on nutritional status in these patients.

OUTLINE: Patients have a small (6 or 8 French) nasogastral feeding tube or enterostomy tube inserted after diagnosis. Peptamen® AF tube feeding is administered via the enteral tube. Tube feedings are started as a continuous drip using an enteral feeding pump with a subsequent steady daily rate increase. Patients receive enteral feeding during courses 1-4 of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly confirmed diagnosis of 1 of the following:

  * Acute myeloid leukemia
  * Myelodysplastic syndromes
  * Sarcoma
  * Any other stage IV solid tumor including:

    * Wilms
    * Neuroblastoma
    * Hepatoblastoma
  * Any primary cancer of the central nervous system including:

    * Cerebellar astrocytoma
    * Medulloblastoma
    * Ependymoma
    * Spine tumors

Exclusion Criteria:

* No contraindication to enteral tube feeding including, but not limited to, any of the following:

  * Gastrointestinal tract dysfunction (i.e., ileus, peritonitis, obstruction)
  * Active sinusitis (can be waived for patients with gastrostomy tubes)
  * Obstructive tumor in the nasopharynx

PRIOR CONCURRENT THERAPY:

* No prior hematopoietic stem cell transplant
* All clinically indicated medications are permitted during the course of the study
* No other concurrent nutritional supplements

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Primary Completion 2008-01 (Estimated); Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Successful administration of enteral feedings via a nasogastric tube for 50% or more of the total nutritional-support days | 50% or more of the total nutritional support days.

SECONDARY OUTCOMES:
Number of patients accepting early insertion of enteral feeding tube for an approximate twelve week period | twelve weeks
Number of times tubes replaced and number of subjects refusing replacement
Grade 3/4 gastrointestinal toxicity associated with enteral support
Complications associated with tube placement
Time to achieve primary goal of meeting 70% of nutritional needs by enteral intake and days maintained at this level | Not indicated
Days of enteral (tube feeding) and total parenteral nutrition
Nutritional status assessment on enrollment in study, beginning of course 1, and end of study period (week 12 or beginning of course 5 chemotherapy | week 12 or beginning course of Chemotherapy
Duration of hospitalization
Need for post-discharge nutritional support

CONTACTS AND LOCATIONS:
Overall Officials: John B. Pietsch, MD, Study Chair — Vanderbilt-Ingram Cancer Center